CLINICAL TRIAL: NCT07373860
Title: Investigation of the Relationship Between Frailty Status and Pain Type, Pain Localization, and GNRI in Individuals Aged 65 Years and Older With Chronic Pain Presenting to a Pain Clinic
Brief Title: Frailty and Chronic Pain Profiles in Patients Aged ≥65 Years
Acronym: F&P
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Assoc. prof., Ankara City Hospital Bilkent
Other Study IDs: TABED-1-25-1637
Record Dates: First submitted 2026-01-15; First posted 2026-01-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Geriatric Pain
Keywords: chronical pain; neuropathic pain; Nociceptive Pain
MeSH Terms: conditions — Neuralgia; Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Chronic Pain Cohort: The Elderly Chronic Pain Cohort consisted of individuals aged 65 years and older who presented to the pain outpatient clinic with complaints of chronic pain and met the study inclusion criteria. All eligible participants were consecutively enrolled during the study period. Frailty status, nutritional risk, and pain-related characteristics were systematically assessed at baseline. Subgroup analyses were performed according to frailty statu

SUMMARY:
The primary aim of this study is to investigate the relationship between frailty status and pain type, pain localization, and the Geriatric Nutritional Risk Index (GNRI) in individuals aged 65 years and older who present to an pain clinic with chronic pain. The secondary aim is to evaluate the level of interaction among these parameters and to contribute to a holistic approach to pain management in older adults.

DETAILED DESCRIPTION:
This study is an observational, cross-sectional investigation to be conducted in individuals aged 65 years and older who present to the algology outpatient clinic with complaints of chronic pain. Participation in the study will be entirely voluntary, and written informed consent will be obtained from all participants. Data collection will be carried out through face-to-face interviews with patients and retrospective review of patient medical records.

Frailty status of the participants will be assessed using the FRAIL Scale, which is widely used in the literature and has proven validity. Alternatively, the Fried Frailty Criteria may be used according to the researcher's preference. Based on these assessments, frailty status will be classified into three categories: robust, prefrail, and frail.

The Geriatric Nutritional Risk Index (GNRI), an objective indicator of nutritional status, will be calculated using participants' serum albumin levels, current body weight, and height according to the following formula:

GNRI = (1.489 × serum albumin [g/L]) + (41.7 × current body weight / ideal body weight).

This score will be analyzed in relation to frailty status to evaluate nutritional risk.

As part of pain assessment, pain intensity will be measured using the Visual Analog Scale (VAS). To determine pain type, the DN4 (Douleur Neuropathique 4) questionnaire and the painDETECT questionnaire, both of which have established validity for neuropathic pain assessment, will be administered. In addition, pain localization will be classified using a pain localization map, and multisite pain involvement will also be recorded.

All collected data will be recorded in encrypted data forms and stored digitally with access restricted to the research team only. Personal identifying information will not be used at any stage of the study, and full compliance with the principles of confidentiality and privacy will be ensured.This study is an observational, cross-sectional investigation to be conducted in individuals aged 65 years and older who present to the algology outpatient clinic with complaints of chronic pain. Participation in the study will be entirely voluntary, and written informed consent will be obtained from all participants. Data collection will be carried out through face-to-face interviews with patients and retrospective review of patient medical records.

Frailty status of the participants will be assessed using the FRAIL Scale, which is widely used in the literature and has proven validity. Alternatively, the Fried Frailty Criteria may be used according to the researcher's preference. Based on these assessments, frailty status will be classified into three categories: robust, prefrail, and frail.

The Geriatric Nutritional Risk Index (GNRI), an objective indicator of nutritional status, will be calculated using participants' serum albumin levels, current body weight, and height according to the following formula:

GNRI = (1.489 × serum albumin [g/L]) + (41.7 × current body weight / ideal body weight).

This score will be analyzed in relation to frailty status to evaluate nutritional risk.

As part of pain assessment, pain intensity will be measured using the Visual Analog Scale (VAS). To determine pain type, the DN4 (Douleur Neuropathique 4) questionnaire and the painDETECT questionnaire, both of which have established validity for neuropathic pain assessment, will be administered. In addition, pain localization will be classified using a pain localization map, and multisite pain involvement will also be recorded.

All collected data will be recorded in encrypted data forms and stored digitally with access restricted to the research team only. Personal identifying information will not be used at any stage of the study, and full compliance with the principles of confidentiality and privacy will be ensured.

ELIGIBILITY:
Inclusion Criteria:

Age 65 years or older Diagnosis of chronic pain (duration > 3 months)

Exclusion Criteria:

Acute pain complaint Pain related to malignancy Severe communication impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who have chronical pain for more than months and older than 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | baseline
  Pain intensity was assessed using the Visual Analog Scale (VAS), ranging from 0 to 10, where higher scores indicate greater pain severity.
primary outcome | baseline
  Frailty was assessed using the Clinical Frailty Scale, ranging from 1 to 9, where higher scores indicate greater frailty.
Primary Outcome Measure | baseline
  Pain type classification (neuropathic, nociceptive, or mixed), assessed at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Saito, Takafumi, et al. "Relationship between chronic pain types (nociceptive and neuropathic-like symptoms) and frailty in community-dwelling Japanese older adults: A cross-sectional study." Journal of Pain Research (2023): 2675-2684.